CLINICAL TRIAL: NCT05869175
Title: Evaluation of the Relationship Between Technology Addiction and Posture Disorder, Balance and Muscle Strength in Preschool Children
Brief Title: Health Problems Caused by Technology Addiction in Preschool Children
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Other Study IDs: Addiction
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Technology Addiction
Keywords: preschool, posture disorder, balance, muscle strength
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Technological products are tools that make human life easier. Among these tools that have become an indispensable part of human life, smart devices, namely smart phones, tablets and computers, have a special place. It is seen that the time spent by both parents and children in the family with smart devices has increased for various reasons. This situation creates effects on the developmental processes of children.

In the literature, it is seen that children and adolescents are more exposed to digital technology. Preschoolers, unlike other children, are in the process of forming healthy habits that will continue to reflect their future quality of life. Incorrect posture in preschool and school-aged children can cause extremely serious health problems in adulthood, if not detected and removed in time. Knowledge of postural control and muscle strength can be important both for identifying children at high risk of falls and injury and for developing fall and injury prevention intervention programs.

More specifically, knowledge of a potential relationship between postural control and muscle strength can assist in tailoring specially designed injury and fall prevention intervention programs.

As a result, with the changing world, the age at which children start using technological devices is gradually decreasing, and as age increases, the duration of device use also increases. Provider, children's exposure to technology will be much longer than adults. There are no studies evaluating the relationship between technology addiction, posture disorder, balance and muscle strength in the preschool period. Generally, research has been done on technology addiction and posture disorder.

The aim of our research is not only to investigate the technology addiction and posture disorder of preschool children, but also to evaluate the relationship between future muscle strength and balance of the posture disorder that may occur.

DETAILED DESCRIPTION:
Technological products are tools that make human life easier. Among these tools that have become an indispensable part of human life, smart devices, namely smart phones, tablets and computers, have a special place. Considering the studies, the age at which children start using technological devices is gradually decreasing and their physical activity is decreasing more because they spend more time with technological devices and are more inactive due to the increase in technology addiction. This situation creates negative effects on the developmental processes of children. Some of these effects are postural disturbance, decreased muscle strength and balance. No study was found that evaluated the relationship between technology addiction, posture disorder, balance and muscle strength in the preschool period. Generally, research has been done on technology addiction and posture disorder.

The aim of this study is not only to investigate the technology addiction and posture disorder of preschool children, but also to evaluate the relationship between future muscle strength and balance of the posture disorder that may occur.

This study can increase the awareness of parents and teachers by detecting health problems such as posture disorder, decrease in muscle strength and balance that may occur due to technology addiction of preschool children, and it can benefit pre-school children to use technology in a beneficial way for their development, both mentally and physically.

ELIGIBILITY:
Inclusion Criteria:

* Having consented to participate in the study by their parents
* Having normal development
* Absence of neurodevelopmental or neuromotor disability

Exclusion Criteria:

* Those who were not approved by their parents to participate in the study.
* Presence of neurodevelopmental or neuromotor disability
* Children with physical or mental disabilities
* Having an orthopedic or metabolic problem

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The preschool period includes 60 children with technology addiction.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Problematic Technology Use scale for Children | First Day
  The scale was published as 26 items. The scale consists of four factors in total, eight items in the Continuity of Use sub-dimension, six items in the second sub-dimension, Resistance to Control, five items in the third sub-dimension, Impact on Development, and seven items in the fourth sub-dimension, Deprivation-Escape.
  In the score calculation of the scale, the statements changing from "I strongly disagree" to "I totally agree" are scored from 1 to 5. The score that can be obtained from the scale varies between 26 and 130. There is no reverse item in the measurement tool. The increase in the score obtained from the measurement tool indicates that the level of problematic technology use of the child increases. The validity and reliability study of the Turkish form of the scale was performed by Ahmet, Onder, and Omer (2022).

SECONDARY OUTCOMES:
New York Posture Analysis | First Day
  Posture changes are observed in 13 different parts of the body, including head, neck, shoulder, back, waist, hip and ankle. According to the results of the observation, five (5) points are given if the person has a correct posture, three (3) points if the posture is moderately impaired, and one (1) point if there is a serious deterioration. The total score obtained as a result of the test varies between 13-65.
Pediatric Balance Scale | First Day
  It includes sitting balance, standing balance, transition from sitting to standing/switching from standing to sitting, transfers, taking a step, reaching forward, reaching down, turning, stepping on a step. It consists of 14 items, each item is scored between 0-4. A score of 0 indicates that he cannot do the instruction, and a score of 4 indicates that he can do it without difficulty. The total score is between 0-56. A low total score indicates a decrease in the balance function.
Muscle Strength | First Day
  After the tests are explained in a way that children can understand, they will be administered with three repetitions of trials and each test will be administered with 15-second rest intervals between tests to prevent fatigue. The isometric contraction force value obtained with the device resistance will be recorded three times and averaged. In all cases, trunk extensors and flexors, bilateral hip flexors, abductors, adductors, extensors, knee extensors and flexors, ankle dorsiflexor and plantarflexor muscle strength values will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Agabek Orunbayev Physiotherapist, Study Chair — Karabuk University; Musa Güneş Msc, Study Director — Karabuk University; Metehan Yana PhD, Principal Investigator — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

REFERENCES:
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Howie EK, Coenen P, Campbell AC, Ranelli S, Straker LM. Head, trunk and arm posture amplitude and variation, muscle activity, sedentariness and physical activity of 3 to 5 year-old children during tablet computer use compared to television watching and toy play. Appl Ergon. 2017 Nov;65:41-50. doi: 10.1016/j.apergo.2017.05.011. Epub 2017 Jun 7. PMID 28802459
- [Background] Hytonen M, Pyykko I, Aalto H, Starck J. Postural control and age. Acta Otolaryngol. 1993 Mar;113(2):119-22. doi: 10.3109/00016489309135778. PMID 8475724
- [Background] Kobel S, Henle L, Laemmle C, Wartha O, Szagun B, Steinacker JM. Intervention Effects of a Kindergarten-Based Health Promotion Programme on Motor Abilities in Early Childhood. Front Public Health. 2020 Jun 30;8:219. doi: 10.3389/fpubh.2020.00219. eCollection 2020. PMID 32695738
- [Background] Taylor NF, Dodd KJ, Graham HK. Test-retest reliability of hand-held dynamometric strength testing in young people with cerebral palsy. Arch Phys Med Rehabil. 2004 Jan;85(1):77-80. doi: 10.1016/s0003-9993(03)00379-4. PMID 14970972
- See also: Problematic Technology Use Scale for Young Children (PTUS-YC): Validity and Reliability Study — https://dergipark.org.tr/en/download/article-file/1609961